CLINICAL TRIAL: NCT01154985
Title: A Phase II Double-Blind, Placebo-Controlled Study of Two Doses of EPA-E in Patients With NASH
Brief Title: Double-Blind, Placebo-Controlled Study of Two Doses of EPA-E in Patients With Non Alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mochida Pharmaceutical Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCH-02-001
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-10

CONDITIONS: Steatohepatitis
Keywords: omega-3 fatty acids; alanine transaminase; triglycerides; lipids; EPA; ethyl-EPA; ethyl icosapentate; Non Alcoholic steatohepatitis; Non Alcoholic fatty liver disease; fatty acids
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): 3x placebo capsules TID
  Interventions: Drug: Placebo capsule
- EPA-E 1800 mg/day (Experimental): 2x EPA-E 300 mg capsules + 1placebo capsule TID
  Interventions: Drug: EPA-E 300 mg capsule
- EPA-E 2700 mg/day (Experimental): 3x EPA-E 300 mg capsules TID
  Interventions: Drug: EPA-E 300 mg capsule

INTERVENTIONS:
Drug: Placebo capsule — 3x Placebo capsules three times a day (TID) for 365 days
  Arms: Placebo
Drug: EPA-E 300 mg capsule — 2x 300 mg capsules + placebo capsule TID for 365 days
  Arms: EPA-E 1800 mg/day
Drug: EPA-E 300 mg capsule — 3x 300 mg capsules TID for 365 days
  Arms: EPA-E 2700 mg/day

SUMMARY:
This is a controlled study to determine the effectiveness and safety of ethyl icosapentate (EPA-E) in the treatment of adult patients with non-alcoholic steatohepatitis (NASH).

DETAILED DESCRIPTION:
This is a phase II, double-blinded, placebo-controlled study to investigate the safety, efficacy, and pharmacokinetic profile of two doses of EPA-E in adult subjects with NASH. Subjects are required to have a liver biopsy with proven NASH in the 6 month period prior to screening. Up to 70 subjects will be enrolled into each treatment arm in a 1:1:1 ratio, for a total of 210 subjects. Subjects will be stratified at randomization by presence or absence of diabetes. Duration of treatment is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite NASH
* Patients with diabetes taking stable doses of anti-diabetic agents are eligible
* No significant concomitant medical illness

Exclusion Criteria:

* Diagnosis of cirrhosis.
* Serum ALT > 300 U/L
* Use of drugs associated with steatohepatitis
* Use of the following anit-NASH agents:

  1. Vitamin E > 60 IU per day
  2. Omega-3-acid ethyl esters or omega-3-polyunsaturated fatty acid (PUFA)-containing supplements > 200 mg per day
  3. Thiazolidinediones (e.g. pioglitazone)
* Use of non-stable doses of the following anti-NASH agents: HMGCoA reductase inhibitors (statins), fibrates, probucol, ezetimibe, ursodiol (UDCA), taurine, betaine, N-acetylcysteine, s-adenosylmethionine (SAM-E), milk thistle, anti-TNF therapies, or probiotics.
* Other liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2010-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (31):
  - Mochida Investigative Site, Dothan, Alabama
  - Mochida Investigative Site, Tucson, Arizona
  - Mochida Investigative Site, Anaheim, California
  - Mochida Investigative Site, Coronado, California
  - Mochida Investigative Site, La Jolla, California
  - Mochida Investigative Site, Los Angeles, California
  - Mochida Investigative Site, San Diego, California
  - Mochida Investigative Site, Littleton, Colorado
  - Mochida Investigative Site, Hialeah, Florida
  - Mochida Investigative Site, Chicago, Illinois
  - Mochida Investigative Site, Lexington, Kentucky
  - Mochida Investigative Site, New Orleans, Louisiana
  - Mochida Investigative Site, Chevy Chase, Maryland
  - Mochida Investigative Site, Detroit, Michigan
  - Mochida Investigative Site, Plymouth, Minnesota
  - Mochida Investigative Site, Jackson, Mississippi
  - Mochida Investigative Site, Tupelo, Mississippi
  - Mochida Investigative Site, Plainview, New York
  - Mochida Investigative Site, Asheville, North Carolina
  - Mochida Investigative Site, Durham, North Carolina
  - Mochida Investigative Site, Cincinnati, Ohio
  - Mochida Investigative Site, Cleveland, Ohio
  - Mochida Investigative Site, Providence, Rhode Island
  - Mochida Investigative Site (2 sites), Germantown, Tennessee
  - Mochida Investigative Site, Nashville, Tennessee
  - Mochida Investigative Site, Houston, Texas
  - Mochida Investigative Site (2 sites), Houston, Texas
  - Mochida Investigative Site, San Antonio, Texas
  - Mochida Investigative Site, Newport News, Virginia
  - Mochida Investigative Site, Richmond, Virginia
  - Mochida Investigative Site, Seattle, Washington
- Mochida Investigative Site, San Juan, Puerto Rico, Puerto Rico

REFERENCES:
- [Derived] Sanyal AJ, Abdelmalek MF, Suzuki A, Cummings OW, Chojkier M; EPE-A Study Group. No significant effects of ethyl-eicosapentanoic acid on histologic features of nonalcoholic steatohepatitis in a phase 2 trial. Gastroenterology. 2014 Aug;147(2):377-84.e1. doi: 10.1053/j.gastro.2014.04.046. Epub 2014 May 9. PMID 24818764

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo: Placebo three times a day (TID) for 365 days
- EPA-E 1800 mg/Day: EPA-E: 600 mg TID for 365 days
- EPA-E 2700 mg/Day: EPA-E: 900 mg TID for 365 days
Period: Overall Study
Arm/Group | Placebo | EPA-E 1800 mg/Day | EPA-E 2700 mg/Day
Started | 75 (Randomized) | 82 (Randomized) | 86 (Randomized)
Full Analysis Set | 75 (Received at least one dose of study medication) | 82 (Received at least one dose of study medication) | 86 (Received at least one dose of study medication)
Valid Biopsy -Baseline and Month 12.5 | 60 | 62 | 68
Efficacy Evaluable Analysis Set | 55 (12-months histological data, no major protocol violations; after minimum 6 months treatment) | 55 (12-months histological data, no major protocol violations; after minimum 6 months treatment) | 64 (12-months histological data, no major protocol violations; after minimum 6 months treatment)
Completed | 58 | 55 | 68
Not Completed | 17 | 27 | 18

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | EPA-E 1800 mg/Day | EPA-E 2700 mg/Day | Total
Number analyzed (Participants) | 75 | 82 | 86 | 243
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 67 | 74 | 80 | 221
  >=65 years | 8 | 8 | 6 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (12.45) | 47.8 (12.48) | 47.8 (11.14) | 48.6 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 48 | 57 | 148
  Male | 32 | 34 | 29 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 15 | 45
  Not Hispanic or Latino | 60 | 67 | 71 | 198
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 2 | 3
  Asian | 3 | 1 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 3 | 3 | 2 | 8
  White | 68 | 77 | 75 | 220
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Histological Response Defined by Change From Baseline in Standardized Scoring of Liver Biopsies
Description: Patient is considered a responder if histological examination shows:
  Composite NAS of <=3 AND no worsening in Fibrosis OR Improvement in NAS by >=2 across at least 2 of the NAS components AND no worsening in fibrosis
  A priori threshold for statistical significance is p<0.05, 1-sided
Time Frame: 12 months
Population: Efficacy Evaluable Analysis Set - All patients in Full Analysis Set who have valid 12-month histological data without major protocol violations, including withdrawn patients with valid 12.5 month histological data after more than 6 months treatment
Measure: Number; unit: participants
Arm/Group | Placebo | EPA-E 1800 mg/Day | EPA-E 2700 mg/Day
Number analyzed (Participants) | 55 | 55 | 64
participants | 18 | 18 | 20
Statistical Analysis 1: Comparison: Placebo vs EPA-E 1800 mg/Day vs EPA-E 2700 mg/Day; Proportion of responders in the EPA-E 1800 mg and 2700 mg groups compared to the proportion of responders in the placebo group compared using the Cochran-Armitage trend test in the Efficacy Evaluable analysis set. P-value less than 5% 1-sided. A total sample size of 210 (70 per arm) was planned to give 80% power for detecting a positive dose-response slope among the 3 treatment arms at 12 months; Test type: Superiority or Other; p = 0.57, Cochran-Armitage trend test

2. Primary Outcome: Alanine Transaminase (ALT) Levels
Description: Mean change from baseline at month 3 analyzed by Analysis of Covariance (ANCOVA) in the efficacy evaluable analysis set with treatment group as a factor and baseline ALT as a covariate. Principal comparisons were the response between;
  1. EPA-E 2700 mg and Placebo groups
  2. EPA-E 1800 mg and Placebo groups
Time Frame: 3 month endpoint
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Placebo | EPA-E 1800 mg/Day | EPA-E 2700 mg/Day
Number analyzed (Participants) | 55 | 55 | 64
U/L | -19.3 (4.61) | -3.0 (4.61) | 2.8 (4.27)
Statistical Analysis 1: Comparison: Placebo vs EPA-E 1800 mg/Day; Least Squares (LS) mean, 95% CI and 2-sided p-value obtained from ANCOVA model with treatment group as a factor and baseline ALT as a covariate. 1,800 mg/day EPA-E treatment group compared to placebo; Test type: Superiority or Other; p = 0.0137, ANCOVA — Two-sided p-values testing for significance was performed within treatment group change from baseline and comparisons between treatment groups. Multiple comparison techniques were not applied
Statistical Analysis 2: Comparison: Placebo vs EPA-E 1800 mg/Day; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 16.2, 95% CI 2-sided [3.4 to 29.1]
Statistical Analysis 3: Comparison: Placebo vs EPA-E 2700 mg/Day; Least Squares (LS) mean, 95% CI and 2-sided p-value obtained from ANCOVA model with treatment group as a factor and baseline ALT as a covariate. 2,700 mg/day EPA-E treatment group compared to placebo; Test type: Superiority or Other; p = 0.0006, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs EPA-E 2700 mg/Day; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; Mean Difference (Final Values) = 22.0, 95% CI 2-sided [9.6 to 34.4]

3. Primary Outcome: Alanine Transaminase (ALT) Levels
Description: Mean change from baseline at month 6 analyzed by Analysis of Covariance (ANCOVA) in the efficacy analysis set with treatment group as a factor and baseline ALT as a covariate. Principal comparisons were the response between;
  1. EPA-E 2700 mg and Placebo groups
  2. EPA-E 1800 mg and Placebo groups
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | EPA-E 1800 mg/Day | EPA-E 2700 mg/Day
Number analyzed (Participants) | 55 | 55 | 64
U/L | -19.1 (4.79) | -9.5 (4.80) | -3.0 (4.45)
Statistical Analysis 1: Comparison: Placebo vs EPA-E 1800 mg/Day; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1592, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs EPA-E 1800 mg/Day; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 9.6, 95% CI 2-sided [-3.8 to 23.0]
Statistical Analysis 3: Comparison: Placebo vs EPA-E 2700 mg/Day; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0153, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs EPA-E 2700 mg/Day; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; Mean Difference (Final Values) = 16.0, 95% CI 2-sided [3.1 to 28.9]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events solicited at each study visit.
Arm/Group | Placebo | EPA-E 1800 mg/Day | EPA-E 2700 mg/Day
Serious Adverse Events (participants affected / at risk) | 4/75 | 8/82 | 5/86
Other Adverse Events (participants affected / at risk) | 71/75 | 65/82 | 74/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | EPA-E 1800 mg/Day (N=82) | EPA-E 2700 mg/Day (N=86)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 2 | 0
pancreatitis relapsing (Gastrointestinal disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 0
Asthenia (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Post procedural pneumonia (Infections and infestations) | 0 | 0 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural hematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Carcinoid tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Transient ischemic attack (Nervous system disorders) | 0 | 2 | 0
Complicated migraine (Nervous system disorders) | 0 | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | EPA-E 1800 mg/Day (N=82) | EPA-E 2700 mg/Day (N=86)
Anaemia (Blood and lymphatic system disorders) | 4 | 3 | 2
Nausea (Gastrointestinal disorders) | 7 | 8 | 16
Diarrhoea (Gastrointestinal disorders) | 13 | 6 | 11
Vomiting (Gastrointestinal disorders) | 4 | 3 | 10
Abdominal pain (Gastrointestinal disorders) | 4 | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3 | 6
Gastroesphageal reflux disease (Gastrointestinal disorders) | 4 | 2 | 4
Fatigue (General disorders) | 6 | 3 | 4
Oedema peripheral (General disorders) | 6 | 3 | 4
Pyrexia (General disorders) | 4 | 2 | 3
Urinary tract infection (Infections and infestations) | 11 | 11 | 8
Nasopharyngitis (Infections and infestations) | 9 | 3 | 6
Sinusitis (Infections and infestations) | 5 | 4 | 7
Gastroenteritis viral (Infections and infestations) | 3 | 2 | 8
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 5
Bronchitis (Infections and infestations) | 5 | 1 | 4
Diverticulitis (Infections and infestations) | 4 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 4 | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 4 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 5
Dizziness (Nervous system disorders) | 4 | 4 | 1
Depression (Psychiatric disorders) | 4 | 4 | 4
Hypertension (Vascular disorders) | 5 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No